CLINICAL TRIAL: NCT04892160
Title: Comparison of Guided Imagery and Virtual Reality (VR) Technology on Patient and Parent Coping and Resource Utilization During Unsedated Procedures
Brief Title: Distracting Through Procedural Pain and Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Northwestern Mutual Foundation (Unknown)
Responsible Party: Principal Investigator, Jennifer Hoag, Associate Professor of Pediatrics, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1110230
Record Dates: First submitted 2021-05-07; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Chronic Illness; Hematologic Malignancy; Bone Marrow Transplant Infection; Oncology; Sickle Cell Disease
Keywords: Procedural Pain; Anxiety; Pediatric; Virtual Reality; Guided Imagery
MeSH Terms: conditions — Chronic Disease; Hematologic Neoplasms; Neoplasms; Anemia, Sickle Cell; Pain, Procedural; Anxiety Disorders | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery First/Virtual Reality Second (Other): Patients will be played a guided imagery experience first during one of the following procedures: port access, dressing changes, and IV sticks. The second scheduled procedure will be the same procedure as the first and occur within 5 to 40 days. At the time of their second procedure, they will receive the virtual reality intervention.
  Interventions: Other: Guided Imagery; Other: Virtual Reality
- Virtual Reality First/Guided Imagery Second (Experimental): Patients will have the VR interactive experience played first during one of the following procedures: port access, dressing changes, and IV sticks. The second scheduled procedure will be the same procedure as the first and occur within 5 to 40 days. At the time of their second procedure, they will receive the guided imagery intervention.
  Interventions: Other: Guided Imagery; Other: Virtual Reality

INTERVENTIONS:
Other: Guided Imagery — Upon completion of study paperwork and 3-5 minutes prior to the nurse entering the room, study personnel will play an audio recording of an underwater guided imagery during one of these procedures: port access, dressing changes, and IV sticks. Guided imagery is an intervention that relies on a patient's imagination to create a sensory experience that utilizes mental images, sounds, smells, tastes, and touch. The guided imagery script used in this study describes an underwater scene and is meant to closely mimic the VR condition with the exception that it will be non-immersive. It will last approximately 15 minutes but can be played again if the procedure lasts longer than 15 minutes. Study personnel will remain in the room to record the time of the procedure, staff number, time in the room, and complete an observational measure of distress.
Other: Virtual Reality — Upon completion of study paperwork and 3-5 minutes prior to the nurse entering the room, study personnel will assist the patient in beginning the VR intervention during one of these procedures: port access, dressing changes, and IV sticks. The VR intervention consists of interactive audio and visual underwater experience. The VR software offers both passive and active gameplay over the course of 15 minutes, which can be repeated. In the passive experience, the software moves patients through an ocean filled with sea creatures and allows them to look around and observe the underwater scene. In the active experience, patients launch balls at the fish. Patients will be encouraged but not required to actively participate; staff will record whether the patient participates in the active portion of the VR program. Study personnel will remain in the room to record the time of the procedure, staff number, time in the room, and complete an observational measure of distress.

SUMMARY:
Children with acute and chronic illness undergo frequent, painful, and distressing procedures. This randomized control trial was used to evaluate the effectiveness of guided imagery (GI) vs virtual reality (VR) on the procedural pain and state anxiety of children and young adults undergoing un-sedated procedures. We explored the role of trait anxiety and pain catastrophizing in intervention response.

DETAILED DESCRIPTION:
Treatment for pediatric cancer and blood disorders can range from several months to several years. During the course of treatment, children often undergo several painful and/or frightening procedures. Common unsedated procedures include needle access of an implanted central venous port (i.e., "port access") prior to receiving chemotherapy; intravenous needle sticks to provide chronic transfusion therapy or treatment for iron overload in patients with sickle cell disease; and weekly changing of the bandage (dressing) around a peripherally inserted central catheter (PICC). These procedures are often distressing to a pediatric patient. As a result, there is an emphasis on the use of non-pharmacologic interventions to manage symptoms of patient pain and anxiety for procedures that do not warrant pharmacologic intervention. There is also ample evidence to suggest that parental coping is associated with child distress, which highlights the need for interventions that have the potential to decrease parental, as well as patient, distress. Interventions that are cost-effective and sustainable are most appealing in the current healthcare environment.

Non-immersive distraction, such as guided imagery, is widely regarded as useful in decreasing pain and anxiety during procedures. Guided imagery is a cognitive strategy that typically involves a staff member describing in detail a situation that is incompatible with the experience of pain and is meant to invoke feelings of calm. It is a commonly used intervention to address procedural distress and, aside from staff time, is free of cost. However, that the more distracting the stimuli, the greater the expenditure of cognitive energy, and the greater reduction in one's capacity to process pain and feel distressed. This leads one to question whether VR, an immersive, interactive technology that can realistically project three-dimensional images, may be more effective than a non-immersive distraction in managing procedure-related pain and distress. VR has been used to assist with procedural distress in several contexts over the past 15 years, including pediatric pain, burn care, dental procedures, and port access. Reviews of VR usage have been generally positive, with most studies suggesting that VR is a feasible and efficacious method of distraction that can reduce patient-reported and objective physiological measures of pain and distress. Effect sizes in the medium to the large range have been found when comparing VR to standard of care and non-immersive distraction (e.g., videogames), have found that subjects using VR distraction for pain showed more improvement than approximately 83% of control subjects. Other sources have highlighted positive patient satisfaction and a low incidence of negative side effects (e.g., motion sickness) when using VR. The cost of VR equipment has decreased over the years, although VR headsets still average $300-500 with additional cost for game controllers and smartphones/game systems. For use within a hospital, the further cost would need to be incurred to reduce the risk of infection for equipment that is shared.

Using a comparative effectiveness model, this project will compare a low-cost, but widely accepted non-immersive distraction intervention (guided imagery) to a higher cost, but very promising immersive intervention (VR) in managing patient pain and anxiety, as well as parent distress. To our knowledge, this is the first time these two interventions will be directly compared. It is also the first time that parental distress will be measured as an outcome of a VR intervention. Hospital resource utilization (staff time, facility usage) will be evaluated as an additional cost/benefit aspect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals being seen by the hematology, oncology, and blood and marrow transplant services.
* English-speaking patients between the ages of 8-25 years that are at least one month post-diagnosis.
* Has one of the three qualifying procedures: port access, dressing changes, and IV sticks.

Exclusion Criteria:

* Patients having identified physical impairments (e.g., blindness, active infection of the skin, history of seizure disorder) that would prevent them from using VR equipment.
* Patients with significant developmental delays that would prevent them from completing required study forms.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
GI vs. VR in patient pain via the Pain Catastrophizing Scale (PCS) | The PCS will be completed by the patient 10 minutes before the first procedure or intervention (i.e., at baseline).
  GI will be compared to VR when it comes to the Pain Catastrophizing Scale for Children (PCS) to identify subgroups that may respond better to one intervention over another. Patient perceptions of pain will be assessed prior to the first procedure using either the child (for patients 8-16 years) or adult (for patients 17+ years) version of the Pain Catastrophizing Scale (PCS). The PCS is a 13-question survey which assesses thoughts and feelings related to pain on a 5 point scale ranging from "not at all" to "extremely."
GI vs. VR in patient pain via the Visual Analogue Scale (VAS) | The VAS will be completed by the patient within 10 minutes after completion of each intervention (i.e., GI and VR intervention).
  GI will be compared to VR when it comes to the Visual Analogue Scale (VAS). This measure is used to assess pain and distress across 6 domains: (1) highest level of pain, (2) average amount of pain, (3) anxiety about pain, (4) unpleasantness of pain, (5) bothersomeness of pain, and (6) time spent thinking about pain. Scores range from 0-100 on each item.
GI vs. VR in patient pain via Children's Emotional Manifestation of Pain Scale (CEMS) | The CEMS will be completed by study staff during each intervention. Study staff will assess the patients through the duration of the procedure and intervention that same day.
  GI will be compared to VR when it comes to the Children's Emotional Manifestation of Pain (CEMS). This observational measure offers an objective way to measure distress during difficult medical experiences. It includes the following domains: anxiety score, facial expression, vocalization, activity, interaction, and level of cooperation.
GI vs. VR in patient anxiety via State Trait Anxiety Inventory - Trait (STAI-T) | The STAI-T will be completed by the patient 10 minutes before the first procedure or intervention (i.e., at baseline).
  GI will be compared to VR when it comes to the State-Trait Anxiety Inventory-Trait (STAI-T) to identify subgroups that may respond better to one intervention over another. This measure is used to assess a patient's trait (underlying or baseline) anxiety. There is a child portion for patients 8-16 years or an adult portion for patients 17+ years.
GI vs. VR in patient anxiety via STAI-State Pre-Intervention | STAI-State will be completed 10 minutes prior to the first and second procedure (GI and VR).
  GI will be compared to VR when it comes to the STAI-State. This assessment is used to assess a patient's state (in the moment) anxiety. There is only one version for all ages.
GI vs. VR in patient anxiety via STAI-State Post-Intervention | STAI-State will be completed 10 minutes after the first and second intervention (GI and VR).
  GI will be compared to VR when it comes to the STAI-State. This assessment is used to assess a patient's state (in the moment) anxiety. There is only one version for all ages.

SECONDARY OUTCOMES:
GI vs. VR in parent distress via PCS-P | The PCS-P will be completed by the caregiver 10 minutes before the first procedure or intervention.
  GI will be compared to VR when it comes to the Pain Catastrophizing Scale for Parents (PCS-P). The PCS-P is a caregiver perspective, that consists of a 13-question survey that assesses thoughts and feelings related to children's pain on a 5 point scale ranging from "not at all" to "extremely."
GI vs. VR in parent distress via Emotional Adjective Survey | The Emotion Adjective Survey will be completed by the caregiver 10 minutes after each intervention.
  GI will be compared to VR when it comes to the Emotion Adjective Survey. The Emotion Adjective Survey is a measure of caregiver distress that asks for a rating of distress across four emotional experiences (worried, upset, anxious, sad).
GI vs VR in hospital resource utilization via Staff Time | The Staff Time log is completed by a member of the study team. It begins once the nursing staff member opens the sterile kit used for the current procedure and ends when the procedure is completed after each intervention.
  GI will be compared to VR when it comes to Staff Time. This tracking log keeps track of the total number and time (minutes) that nursing staff spend in the patient room during each procedure.
GI vs VR in hospital resource utilization via Procedure Time | The Procedure Time log is completed by a member of the study team. The time begins once the nursing staff member opens the sterile kit used for the current procedure and ends when the procedure is completed/
  GI will be compared to VR when it comes to Procedure Time. This tracking log keeps track of the total time that it takes nursing to complete the procedure.
Nurse Feasibility and Acceptability | The Nurse Feasibility and Acceptability survey will be completed within one day following completion of each intervention.
  Nurses will complete a brief measure assessing feasibility, acceptability, and expectations for success.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hoag, PhD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Children's Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
We will only share de-identified data for researchers who would like to do a secondary analysis.
Supporting Information: Study Protocol, SAP
Time Frame: We will share study documents once the manuscript has been published.
Access Criteria: A researcher who would like to use our data has to contact and get permission from the PI, Jennifer Hoag, PhD.

REFERENCES:
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Blount, R.L., Zempsky, W.T., Jaaniste, T., Evans, S., Cohen, L.L., Devine, K.A., & Zeltzer, L.K. (2009). Management of pediatric pain and distress due to medical procedures. In M.C. Roberts & R.G. Steele (Eds.), Handbook of Pediatric Psychology (pp. 171-188), New York: The Guilford Press.
- [Background] Dahlquist LM, McKenna KD, Jones KK, Dillinger L, Weiss KE, Ackerman CS. Active and passive distraction using a head-mounted display helmet: effects on cold pressor pain in children. Health Psychol. 2007 Nov;26(6):794-801. doi: 10.1037/0278-6133.26.6.794. PMID 18020853
- [Background] Das DA, Grimmer KA, Sparnon AL, McRae SE, Thomas BH. The efficacy of playing a virtual reality game in modulating pain for children with acute burn injuries: a randomized controlled trial [ISRCTN87413556]. BMC Pediatr. 2005 Mar 3;5(1):1. doi: 10.1186/1471-2431-5-1. PMID 15745448
- [Background] Deraney J, Davis M, Evers HB, German K, Hamill JC, Karas-Irwin BS, Mazzer MC, Shaw RE. Drumming Effect on Anxiety. Arch Psychiatr Nurs. 2017 Oct;31(5):528-529. doi: 10.1016/j.apnu.2017.05.001. Epub 2017 May 13. No abstract available. PMID 28927519
- [Background] Gershon J, Zimand E, Lemos R, Rothbaum BO, Hodges L. Use of virtual reality as a distractor for painful procedures in a patient with pediatric cancer: a case study. Cyberpsychol Behav. 2003 Dec;6(6):657-61. doi: 10.1089/109493103322725450. PMID 14756933
- [Background] Gershon J, Zimand E, Pickering M, Rothbaum BO, Hodges L. A pilot and feasibility study of virtual reality as a distraction for children with cancer. J Am Acad Child Adolesc Psychiatry. 2004 Oct;43(10):1243-9. doi: 10.1097/01.chi.0000135621.23145.05. PMID 15381891
- [Background] Gold, J. I., Kant, A. J., & Kim, S. H. (2005, December). Virtual anesthesia: the use of virtual reality for pain distraction during acute medical interventions. In Seminars in Anesthesia, Perioperative Medicine and Pain (Vol. 24, No. 4, pp. 203-210). WB Saunders.
- [Background] Hoffman HG, Doctor JN, Patterson DR, Carrougher GJ, Furness TA 3rd. Virtual reality as an adjunctive pain control during burn wound care in adolescent patients. Pain. 2000 Mar;85(1-2):305-9. doi: 10.1016/s0304-3959(99)00275-4. PMID 10692634
- [Background] Jeffs D, Dorman D, Brown S, Files A, Graves T, Kirk E, Meredith-Neve S, Sanders J, White B, Swearingen CJ. Effect of virtual reality on adolescent pain during burn wound care. J Burn Care Res. 2014 Sep-Oct;35(5):395-408. doi: 10.1097/BCR.0000000000000019. PMID 24823326
- [Background] Kazak AE, Penati B, Brophy P, Himelstein B. Pharmacologic and psychologic interventions for procedural pain. Pediatrics. 1998 Jul;102(1 Pt 1):59-66. doi: 10.1542/peds.102.1.59. PMID 9651414
- [Background] Koller D, Goldman RD. Distraction techniques for children undergoing procedures: a critical review of pediatric research. J Pediatr Nurs. 2012 Dec;27(6):652-81. doi: 10.1016/j.pedn.2011.08.001. Epub 2011 Oct 13. PMID 21925588
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654
- [Background] Nilsson S, Finnstrom B, Kokinsky E, Enskar K. The use of Virtual Reality for needle-related procedural pain and distress in children and adolescents in a paediatric oncology unit. Eur J Oncol Nurs. 2009 Apr;13(2):102-9. doi: 10.1016/j.ejon.2009.01.003. Epub 2009 Feb 20. PMID 19230769
- [Background] Powers SW. Empirically supported treatments in pediatric psychology: procedure-related pain. J Pediatr Psychol. 1999 Apr;24(2):131-45. doi: 10.1093/jpepsy/24.2.131. PMID 10361392
- [Background] Sander Wint S, Eshelman D, Steele J, Guzzetta CE. Effects of distraction using virtual reality glasses during lumbar punctures in adolescents with cancer. Oncol Nurs Forum. 2002 Jan-Feb;29(1):E8-E15. doi: 10.1188/02.ONF.E8-E15. PMID 11845217
- [Background] Schneider SM, Workman ML. Effects of virtual reality on symptom distress in children receiving chemotherapy. Cyberpsychol Behav. 1999;2(2):125-34. doi: 10.1089/cpb.1999.2.125. PMID 19178248
- [Background] Schneider SM, Prince-Paul M, Allen MJ, Silverman P, Talaba D. Virtual reality as a distraction intervention for women receiving chemotherapy. Oncol Nurs Forum. 2004 Jan-Feb;31(1):81-8. doi: 10.1188/04.ONF.81-88. PMID 14722591
- [Background] Sharar SR, Carrougher GJ, Nakamura D, Hoffman HG, Blough DK, Patterson DR. Factors influencing the efficacy of virtual reality distraction analgesia during postburn physical therapy: preliminary results from 3 ongoing studies. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S43-9. doi: 10.1016/j.apmr.2007.09.004. PMID 18036981
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Uman LS, Chambers CT, McGrath PJ, Kisely S. A systematic review of randomized controlled trials examining psychological interventions for needle-related procedural pain and distress in children and adolescents: an abbreviated cochrane review. J Pediatr Psychol. 2008 Sep;33(8):842-54. doi: 10.1093/jpepsy/jsn031. Epub 2008 Apr 2. PMID 18387963
- [Background] Windich-Biermeier A, Sjoberg I, Dale JC, Eshelman D, Guzzetta CE. Effects of distraction on pain, fear, and distress during venous port access and venipuncture in children and adolescents with cancer. J Pediatr Oncol Nurs. 2007 Jan-Feb;24(1):8-19. doi: 10.1177/1043454206296018. PMID 17185397
- [Background] Wismeijer AA, Vingerhoets AJ. The use of virtual reality and audiovisual eyeglass systems as adjunct analgesic techniques: a review of the literature. Ann Behav Med. 2005 Dec;30(3):268-78. doi: 10.1207/s15324796abm3003_11. PMID 16336078
- [Background] Wolitzky, K., Fivush, R., Zimand, E., Hodges, L., & Rothbaum, B. O. (2005). Effectiveness of virtual reality distraction during a painful medical procedure in pediatric oncology patients. Psychology and health, 20(6), 817-824.
- [Background] Zernikow B, Meyerhoff U, Michel E, Wiesel T, Hasan C, Janssen G, Kuhn N, Kontny U, Fengler R, Gortitz I, Andler W. Pain in pediatric oncology--children's and parents' perspectives. Eur J Pain. 2005 Aug;9(4):395-406. doi: 10.1016/j.ejpain.2004.09.008. PMID 15979020
- [Derived] Hoag JA, Karst J, Bingen K, Palou-Torres A, Yan K. Distracting Through Procedural Pain and Distress Using Virtual Reality and Guided Imagery in Pediatric, Adolescent, and Young Adult Patients: Randomized Controlled Trial. J Med Internet Res. 2022 Apr 18;24(4):e30260. doi: 10.2196/30260. PMID 35436209